CLINICAL TRIAL: NCT01028833
Title: Effects of Power Mobility on the Development and Function of Young Children With Severe Motor Impairments
Brief Title: Effects of Power Mobility on Young Children With Severe Motor Impairments
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2480
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Cerebral Palsy; Arthrogryposis; Spinal Muscular Atrophy; Other Central Nervous System or Musculoskeletal Disorders
Keywords: power wheelchairs; power mobility; young children
MeSH Terms: conditions — Cerebral Palsy; Arthrogryposis; Muscular Atrophy, Spinal; Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Power mobility (Experimental): Intervention included provision of power wheelchair and power mobility training program. Project staff will use structured power mobility training program to teach the children to use the power mobility devices. Project staff will schedule 1-hour sessions with each family 3 times per week for the first month of the project and will decrease in the following manner as the child becomes proficient and develops basic wheelchair maneuvering skills: two one-hour session per week for 4 weeks; one one-hour session per week for 4 weeks; two one-hour sessions per month for 4 weeks; one one-hour session per month for the remainder of the study.
  Interventions: Other: Power mobility
- Control (No Intervention): Children in the control group will not receive any additional intervention, but will continue to receive the early intervention or other services they were receiving prior to enrollment in this study.

INTERVENTIONS:
Other: Power mobility — Project staff will use structured power mobility training program to teach the children to use the power mobility devices. Project staff will schedule 1-hour sessions with each family 3 times per week for the first month of the project and will decrease in the following manner as the child becomes proficient and develops basic wheelchair maneuvering skills: two one-hour session per week for 4 weeks; one one-hour session per week for 4 weeks; two one-hour sessions per month for 4 weeks; one one-hour session per month for the remainder of the study.
  Arms: Power mobility

SUMMARY:
The purpose this study is to determine the effects of power mobility on the development and function of young children of young children whose severe physical disabilities limit their exploratory behaviors and may unnecessarily restrict their cognitive, communication, and social-emotional development.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 14- and 30-months of age
* Must have clinical diagnosis of a motor impairment that prevents functional independent mobility
* Must have adequate vision and hearing to use power mobility device safely
* Must have cognitive abilities equivalent to a 12-month level or alertness and interest in the environment that suggests a trial of power mobility is warranted

Ages: 14 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2008-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Merrill-Palmer-Revised | Entry, 6-months, and 12-months
Pediatric Evaluation of Disability Inventory | Entry, 6-months, 12-months

SECONDARY OUTCOMES:
Child Health Status | Entry
Two-position object permanence test | Entry, 6 months, 12 months
Nonspeech Test | Entry, 6 month, 12 months
Home Observation Measure of the Environment | Entry, 6 months, 12 months
Parenting Stress Inventory | Entry, 6 months, 12 months
Center for Epidemiologic Studies Depression Scale (CES-D) | Entry, 6 months, 12 months
Hollingshead Scale | Entry

CONTACTS AND LOCATIONS:
Overall Officials: Maria A. Jones, PT, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Department of Rehabilitation Sciences, Lee Mitchener Tolbert Center for Develompental Disabilities, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Derived] Mockler SR, McEwen IR, Jones MA. Retrospective Analysis of Predictors of Proficient Power Mobility in Young Children With Severe Motor Impairments. Arch Phys Med Rehabil. 2017 Oct;98(10):2034-2041. doi: 10.1016/j.apmr.2017.05.028. Epub 2017 Jul 5. PMID 28688787